Official Title: A Comparison of Lidocaine, Esmolol, and Placebo Without Use of a Tourniquet for

Relieving Pain From Intravenous Administration of Propofol

NCT04356352

IRB-Approved Date: 11/30/22



Department/Section of Anesthesiology

## <u>A COMPARISON OF LIDOCAINE, ESMOLOL AND PLACEBO WITHOUT USE</u> <u>OF A TOURNIQUET FOR RELIEVING PAIN FROM INTRAVENOUS</u> ADMINISTRATION OF PROPOFOL

Informed Consent Form to Participate in Research Michael Norton, MD, Principal Investigator

#### **SUMMARY**

You are invited to participate in a research study. The purpose of this research is to determine whether lidocaine or esmolol helps to eliminate pain from the injection of propofol that is administered as part of your anesthesia for your procedure when compared to not receiving any numbing medicine at all to help eliminate this injection pain. You are invited to be in this study because you are scheduled to have surgery and will be going to sleep for your procedure. These medications are normally administered to put you to sleep.

Participation in this study will involve your discussing this research study with your anesthesia team as part of the process called informed consent. On the day of your surgery you will be randomized like the flip of a coin to receive one of 3 potential treatments to see how well they prevent the pain or discomfort from the injection of the medication called propofol that is being used to put you to sleep. All research studies involve some risks. A risk to this study that you should be aware of are the risks of receiving the lidocaine and the esmolol. These will be discussed in further detail later in this form. There is the possibility that you may benefit from participation in this study if it demonstrates that one medication works better than the other.

Your participation in this study is voluntary. You do not have to participate in this study if you do not want to. There may be other choices available to you. Some other choices may include receiving the numbing medication You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. The person in charge of this study is Dr. Michael Norton. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study please contact the principal investigator at

If you have any questions, suggestions or concerns about your rights as a volunteer in this research, contact the Institutional Review Board at Advocate at Wake Forest at ...


Adult Consent Form



#### Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you are going to have a surgical procedure and will be receiving propofol in order to put you to sleep for your surgery (also called general anesthesia) Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine whether the active medications of lidocaine or esmolol is more effective when compared to placebo, which is like sugar water and contains no active medication, at preventing the discomfort of receiving propofol when it is being used to put you to sleep for your surgery.

Lidocaine has been approved by the US Food and Drug Administration (FDA) as its use as a local anesthetic (or numbing medication). Esmolol has been approved by the US Food and Drug Administration (FDA) but it has not been approved for use as a local anesthetic to be used under these circumstances.

In this study lidocaine and esmolol will be compared to placebo. A placebo is a substance, like a sugar pill, that is not thought to have any effect on your disease or condition. In this study you will either receive one of the active study medications, lidocaine or esmolol, or placebo which is not active. Placebos are used in research studies to see if the drug being studied really does have an effect.

#### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

150 people at Wake Forest Baptist Medical Center will take part in this study.

#### WHAT IS INVOLVED IN THE STUDY?

You will be randomized into one of the study groups described below. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have a one in three chance of being placed in any group.

You nor your anesthesia provider (the nurse anesthetist or anesthesia resident assisting in your care) will not know which drug you are receiving. Your attending anesthesiologist will know the drug you are receiving. This is done so that a fair evaluation of results can be made. This information is available to the researchers if needed in an emergency.

If you take part in this study, you will arrive at the surgery center and be admitted as you to the holding room in preparation for your surgery as you normally would. After you are admitted you will be randomized to receive either lidocaine, esmolol, or placebo as part of your surgical


Adult Consent Form



medications. This will be administered in the operating room within 30 seconds of your receiving the initial dose of propofol. After the administration of the study medication and propofol, you will be asked to provide a pain score based on how the medication felt as it was given through your IV. You will be asked to provide a number on a scale of 0-3, with 0 being no pain, 1 is mild pain, 2 is moderate pain, and 3 being severe pain. You will then receive the remaining propofol to put you to sleep for your surgery. The anesthesia staff will monitor your blood pressure, heart rate, and oxygen saturation as would be done whether you participate in this research study or not.

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for the duration of your surgical procedure. You can stop participating at any time.

#### WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. Risks and side effects related to the use of the study medications are as follows:

Lidocaine: Potential side effects of receiving lidocaine as a local anesthetic include:

- Nausea (uncommon and mild)
- Dizziness (uncommon and mild)
- Numbness in places where medication is applied (common as this is a local anesthetic and mild)
- Redness or itching where medication is injected (common and mild)

These side effects last less than 30 minutes after injection. There is also remote chance of bruising (due to the needle piercing the skin and varies on length of time it is present based on each individual.

Esmolol: This drug is approved to treat irregular heartbeat or high blood pressure. When Esmolol is given for these conditions it is used at a higher dose and over a longer period of time than as will be given to you in this study. When used as approved, the side effects of Esmolol are:

- Low blood pressure (common and mild)
- Nausea (common and mild)
- Sleepiness (common and mild)
- Confusion (common and mild)
- Anxiety (common and mild)
- Headaches (common and mild)

These side effects are generally temporary because esmolol is a short-acting medication (the effects of the drug do not last long in the body).

We do not know the side effects of using Esmolol as a local anesthetic in preventing pain along

Page **3** of **8**Adult Consent Form



with propofol. Because of this, you will be closely monitored for any side effects that may occur.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other risks that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

If you are randomized to receive a placebo, you may experience more discomfort from the propofol being administered than you would should you receive either lidocaine or esmolol.

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

In previous studies both lidocaine and esmolol have been shown to decrease the injection site pain associated with using propofol as your anesthesia medication to put you to sleep for your procedure. If you agree to take part in this study, you may or may not have decreased injection site pain when you are being put to sleep. We also hope the information learned from this study will benefit other people in the future by showing that using one of these medications works better than the other one in helping to alleviate the discomfort of the administration of the propofol.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options: having your surgery and receiving the normal medications as would any other surgery patient, which may include the use of one of these medications to help alleviate the discomfort of receiving the propofol to put you to sleep for your surgery. You could be treated with either lidocaine or esmolol to help eliminate the discomfort of the propofol administration even if you do not take part in the study.

#### WHAT ARE THE COSTS?

All study costs, including any study medications and procedures related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

#### WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed


Adult Consent Form



unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

#### WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the Department of Anesthesiology, Wake Forest University Health Sciences to cover the costs of the study medications being used. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

### WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Michael Norton at during regular business hours, or after hours.

#### WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any information we collect from you or your medical record about your health or behaviors is considered <u>Protected Health Information</u>. If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study may be placed in your medical record, and may be used to help treat

Page **5** of **8**Adult Consent Form



you, arrange payment for your care, or assist with Medical Center operations. We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the participant's original medical record for verification of clinical trial procedures or data, without violating confidentiality of the participant and to the extent permitted by other applicable laws. If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules. Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for at least six years after the study is finished. After that the research information will be destroyed.

You can tell Dr. Norton that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.


Adult Consent Form



By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

#### WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is shown it would be in your best medical interest, your condition indicates it would be best if you did not participate, you have an unexpected reaction, or other indication. Information that identifies you may be removed from the data or specimens that are collected as part of this study and could be used for future research or shared with others without additional consent.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS? For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Michael Norton at or after hours. The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at or the Research Subject Advocate at Subject Advocate a

#### SIGNATURES

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to


Adult Consent Form



ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|-------------------------------------|-------|-------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |